CLINICAL TRIAL: NCT01384058
Title: The Effect of Ezetimibe 10 mg, Simvastatin 20 mg and the Combination of Simvastatin 20 mg Plus 10 mg Ezetimibe on Low Density Lipoprotein (LDL)-Subfractions in Patients With Type 2 Diabetes
Brief Title: Effect of Ezetimibe or Simvastatin or Both on Low Densitiy Lipoprotein -Subfractions in Patients With Type 2 Diabetes
Acronym: EZE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: Essex Pharma GmbH (Industry)
Responsible Party: Principal Investigator, Karl Winkler, MD, Prof. Dr. med., Kommissarischer Ärztlicher Direktor, University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 442006; 2006-005906-30 (EudraCT Number)
Record Dates: First submitted 2011-06-23; First posted 2011-06-28 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Diabetes Mellitus Type 2; Hypercholesterolemia
Keywords: atherogenic lipoprotein; cardiovascular disease; coronary artery disease; type 2 diabetes; small, dense LDL
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypercholesterolemia; Cardiovascular Diseases; Coronary Artery Disease; Cerebral Palsy | interventions — Ezetimibe; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ezetimibe 10mg/d (Active Comparator): intake of ezetimibe 10mg per day for six weeks after wash-out
  Interventions: Drug: ezetimibe
- Simvastatin 20 mg per day (Active Comparator): intake of simvastatin 20 mg per day for six weeks after wash-out
  Interventions: Drug: simvastatin
- Ezetimibe 10 mg/d and Simvastatin 20mg/d (Active Comparator): intake of ezetimibe 10 mg and simvastatin 20 mg per day for six weeks after wash-out
  Interventions: Drug: Ezetimibe 10/Simvastatin 20

INTERVENTIONS:
Drug: ezetimibe — ezetimibe 10 mg per day for six weeks
  Other Names: Ezetrol 10 mg
  Arms: Ezetimibe 10mg/d
Drug: simvastatin — Simvastatin 20 mg per day for six weeks
  Other Names: Zocor MSD
  Arms: Simvastatin 20 mg per day
Drug: Ezetimibe 10/Simvastatin 20 — Ezetimibe 10mg/Simvastatin 20mg per day for six weeks
  Other Names: Inegy 10/20
  Arms: Ezetimibe 10 mg/d and Simvastatin 20mg/d

SUMMARY:
It is of interest how ezetimibe alone or in combination with statin may influence atherogenic dense Low Density Lipoprotein (dLDL) in patients with type 2 diabetes mellitus. The primary objective of this study will be whether there is a change of the concentrations of Apolipoprotein B (ApoB) in dLDL from baseline in each of the 3 treatment groups.

DETAILED DESCRIPTION:
The selective cholesterol resorption inhibitor ezetimibe belongs to a new class of cholesterol lowering drugs. It is of interest how ezetimibe alone or in combination with statin may influence atherogenic dense Low Density Lipoprotein (dLDL) in patients with type 2 diabetes mellitus.

The primary objective of this study will be whether there is a change of the concentrations of Apolipoprotein B (ApoB) in dLDL from baseline in each of the 3 treatment groups. The comparison between treatment groups is exploratory due to insufficient power to detect any change between treatments.

ELIGIBILITY:
Inclusion Criteria:

* men > 18 and ≤ 75 years
* post-menopausal women ≤ 75 years (follicle stimulating hormone (FSH) >30 mIU/ml, women > 60 years FSH > 20 mIU/ml )
* well controlled diabetes mellitus type II (glycohaemoglobin ≤ 8,0 %)
* LDL-cholesterol ≤ 160 mg/dl
* LDL-subfractions: concentration of apoB-100 in dLDL (LDL-5 und LDL-6) > 25 mg/dl
* written informed consent

Exclusion Criteria:

* participation in a clinical trial within the last 30 d before screening- visit
* patient is unable to give written informed consent
* Body mass index <15 kg/m² and > 35 kg/m²
* clinical atherosclerotic disease (coronary heart disease, peripheral artery disease, carotid artery disease)
* malignoma
* uncontrolled arterial hypertension (>160/>100 mmHg)
* clinically relevant disease of liver and/or kidneys
* clinically relevant endocrinally or hematologic problems
* allergy to study medication (Ezetimibe and/or Simvastatin)
* alcohol- or drug abuse
* laboratory: alanine aminotransferase, aspartate aminotransferase, total bilirubin > 3 x ULN, creatine kinase > 5 x ULN
* Concurrent treatment with potent CYP3A4-inhibitors (e.g. itraconazole, ketoconazole, HIV-protease-inhibitors, erythromycin, clarithromycin, telithromycin und nefazodone)
* other relevant diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-11; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change of the concentration of apolipoprotein B (ApoB) in dense Low Densitiy Lipoprotein (dLDL) from baseline with ezetimibe, simvastatin or the combination of both drugs | baseline and 6 weeks
  multicentre, randomized, open-label study investigation in 6-week effect of ezetimibe (10mg/d), simvastatin (20mg/d) or combination of ezetimibe 10mg/simvastatin 20mg/d on concentrations of dLDL separated by preparative gradient ultracentrifugation in patients with type 2 diabetes.

SECONDARY OUTCOMES:
Change of the concentrations of Total Cholesterol | baseline and 6 weeks
Change of the concentrations of Low Densitiy Lipoprotein (LDL) -Cholesterol | baseline and 6 weeks
Change of the concentrations of High Density Lipoprotein (HDL) -Cholesterol | baseline and 6 weeks
Change of the concentrations of triglycerides | baseline and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karl Winkler, MD, Principal Investigator — University Hospital Freiburg
Locations (2):
- Germany (2):
  - Institut für Stoffwechselforschung, Frankfurt, Germany
  - Stephan Jacob, MD, Villingen-Schwenningen, Germany

REFERENCES:
- [Background] Haffner SM, Lehto S, Ronnemaa T, Pyorala K, Laakso M. Mortality from coronary heart disease in subjects with type 2 diabetes and in nondiabetic subjects with and without prior myocardial infarction. N Engl J Med. 1998 Jul 23;339(4):229-34. doi: 10.1056/NEJM199807233390404. PMID 9673301
- [Background] Reaven GM, Chen YD, Jeppesen J, Maheux P, Krauss RM. Insulin resistance and hyperinsulinemia in individuals with small, dense low density lipoprotein particles. J Clin Invest. 1993 Jul;92(1):141-6. doi: 10.1172/JCI116541. PMID 8325978
- [Background] Austin MA, Edwards KL. Small, dense low density lipoproteins, the insulin resistance syndrome and noninsulin-dependent diabetes. Curr Opin Lipidol. 1996 Jun;7(3):167-71. doi: 10.1097/00041433-199606000-00010. PMID 8818515
- [Background] Winkler K, Abletshauser C, Hoffmann MM, Friedrich I, Baumstark MW, Wieland H, Marz W. Effect of fluvastatin slow-release on low density lipoprotein (LDL) subfractions in patients with type 2 diabetes mellitus: baseline LDL profile determines specific mode of action. J Clin Endocrinol Metab. 2002 Dec;87(12):5485-90. doi: 10.1210/jc.2002-020370. PMID 12466341
- [Background] Austin MA, King MC, Vranizan KM, Krauss RM. Atherogenic lipoprotein phenotype. A proposed genetic marker for coronary heart disease risk. Circulation. 1990 Aug;82(2):495-506. doi: 10.1161/01.cir.82.2.495. PMID 2372896
- [Background] Nigon F, Lesnik P, Rouis M, Chapman MJ. Discrete subspecies of human low density lipoproteins are heterogeneous in their interaction with the cellular LDL receptor. J Lipid Res. 1991 Nov;32(11):1741-53. PMID 1770294
- [Background] Dejager S, Bruckert E, Chapman MJ. Dense low density lipoprotein subspecies with diminished oxidative resistance predominate in combined hyperlipidemia. J Lipid Res. 1993 Feb;34(2):295-308. PMID 8429263
- [Background] Anber V, Griffin BA, McConnell M, Packard CJ, Shepherd J. Influence of plasma lipid and LDL-subfraction profile on the interaction between low density lipoprotein with human arterial wall proteoglycans. Atherosclerosis. 1996 Aug 2;124(2):261-71. doi: 10.1016/0021-9150(96)05842-x. PMID 8830938
- [Background] Nordestgaard BG, Nielsen LB. Atherosclerosis and arterial influx of lipoproteins. Curr Opin Lipidol. 1994 Aug;5(4):252-7. doi: 10.1097/00041433-199408000-00002. PMID 7981955
- [Background] Griffin BA, Freeman DJ, Tait GW, Thomson J, Caslake MJ, Packard CJ, Shepherd J. Role of plasma triglyceride in the regulation of plasma low density lipoprotein (LDL) subfractions: relative contribution of small, dense LDL to coronary heart disease risk. Atherosclerosis. 1994 Apr;106(2):241-53. doi: 10.1016/0021-9150(94)90129-5. PMID 8060384
- [Background] Gardner CD, Fortmann SP, Krauss RM. Association of small low-density lipoprotein particles with the incidence of coronary artery disease in men and women. JAMA. 1996 Sep 18;276(11):875-81. PMID 8782636
- [Background] Stampfer MJ, Krauss RM, Ma J, Blanche PJ, Holl LG, Sacks FM, Hennekens CH. A prospective study of triglyceride level, low-density lipoprotein particle diameter, and risk of myocardial infarction. JAMA. 1996 Sep 18;276(11):882-8. PMID 8782637
- [Background] Lamarche B, Tchernof A, Moorjani S, Cantin B, Dagenais GR, Lupien PJ, Despres JP. Small, dense low-density lipoprotein particles as a predictor of the risk of ischemic heart disease in men. Prospective results from the Quebec Cardiovascular Study. Circulation. 1997 Jan 7;95(1):69-75. doi: 10.1161/01.cir.95.1.69. PMID 8994419
- [Background] Berneis KK, Krauss RM. Metabolic origins and clinical significance of LDL heterogeneity. J Lipid Res. 2002 Sep;43(9):1363-79. doi: 10.1194/jlr.r200004-jlr200. PMID 12235168
- [Background] Blake GJ, Otvos JD, Rifai N, Ridker PM. Low-density lipoprotein particle concentration and size as determined by nuclear magnetic resonance spectroscopy as predictors of cardiovascular disease in women. Circulation. 2002 Oct 8;106(15):1930-7. doi: 10.1161/01.cir.0000033222.75187.b9. PMID 12370215
- [Background] ALTSCHUL R, HOFFER A, STEPHEN JD. Influence of nicotinic acid on serum cholesterol in man. Arch Biochem Biophys. 1955 Feb;54(2):558-9. doi: 10.1016/0003-9861(55)90070-9. No abstract available. PMID 14350806
- [Background] Charman RC, Matthews LB, Braeuler C. Nicotinic acid in the treatment of hypercholesterolemia. A long term study. Angiology. 1972 Jan;23(1):29-35. doi: 10.1177/000331977202300105. No abstract available. PMID 5009984
- [Background] DiPalma JR, Thayer WS. Use of niacin as a drug. Annu Rev Nutr. 1991;11:169-87. doi: 10.1146/annurev.nu.11.070191.001125. No abstract available. PMID 1832551
- [Background] Winkler K, Weltzien P, Friedrich I, Schmitz H, Nickell HH, Hauck P, Hoffmann MM, Baumstark MW, Wieland H, Marz W. Qualitative effect of fenofibrate and quantitative effect of atorvastatin on LDL profile in combined hyperlipidemia with dense LDL. Exp Clin Endocrinol Diabetes. 2004 May;112(5):241-7. doi: 10.1055/s-2004-817970. PMID 15146369
- [Background] Winkler K, Friedrich I, Baumstark MW, Wieland H, März W 2002 Pioglitazone reduces atherogenic dense low density lipoprotein (LDL) particles in patients with type 2 diabetes mellitus. Br J Diabetes Vasc Dis 2:143-148
- [Background] Winkler K, Konrad T, Fullert S, Friedrich I, Destani R, Baumstark MW, Krebs K, Wieland H, Marz W. Pioglitazone reduces atherogenic dense LDL particles in nondiabetic patients with arterial hypertension: a double-blind, placebo-controlled study. Diabetes Care. 2003 Sep;26(9):2588-94. doi: 10.2337/diacare.26.9.2588. PMID 12941723
- [Derived] Winkler K, Jacob S, Muller-Schewe T, Hoffmann MM, Konrad T. Ezetimibe alone and in combination lowers the concentration of small, dense low-density lipoproteins in type 2 diabetes mellitus. Atherosclerosis. 2012 Jan;220(1):189-93. doi: 10.1016/j.atherosclerosis.2011.10.043. Epub 2011 Nov 9. PMID 22115011